CLINICAL TRIAL: NCT05801432
Title: Diabetes Follow-up Study for REduction of cardiovAscular outcoMes: a Coronary Computed Tomographic Angiography Cohort Study
Brief Title: A Study to Evaluate Coronary Atherosclerosis in Patients With Diabetes Mellitus
Acronym: DREAM-CCTA
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Seung-Whan Lee, M.D., Ph.D., Part of cardiology, Principal Investigator, associate professor, Asan Medical Center
Other Study IDs: 2021-0759
Record Dates: First submitted 2023-03-22; First posted 2023-04-06 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the natural history of coronary atherosclerosis development and progression over time by CCTA and to identify risk factors attributable to the development of coronary atherosclerosis in a Korean DM population.

DETAILED DESCRIPTION:
Patients with diabetes mellitus, who underwent initial CCTA (coronary computed tomographic angiography) at the Diabetes Center of the Asan Medical Center between February 2008 and June 2012, will be evaluated for inclusion in the study. All DREAM-CCTA study patients will undergo follow-up CCTA based on order from their primary physician. CCTA and demographic data, medical history, cardiovascular risk factors, and laboratory data was collected in case report forms at the time of the initial CCTA and at the time of follow-up CCTA.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Asymptomatic patients with type 2 DM who had undergone initial CCTA evaluation at the Diabetes Center of the Asan Medical Center between February 2008 and June 2012
* Willing and able to provide informed written consent

Exclusion Criteria:

* Blood test results that the Creatinine level exceeds 1.5 mg/dL
* A person with a history of anaphylaxis or allergic shock associated with a contrast medium
* Pregnant women
* Unable to undergo follow-up CCTA
* Uninterpretable CCTA

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 511 consecutive asymptomatic patients with type 2 DM, who had undergone initial CCTA evaluation at the Diabetes Center of the Asan Medical Center between February 2008 and June 2012, will be screened for enrollment in this study. A member of research team should review the patients' medical history for eligibility. If all eligibility criteria are met and written informed consent is provided, the patient may be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 511 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in coronary atherosclerosis detected by initial and follow-up CCTA | about 10 years after first CCTA
  the natural history of coronary atherosclerotic plaque development and progression over time by CCTA

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No